CLINICAL TRIAL: NCT00612222
Title: Phase II Study of Metastatic Melanoma Using Lymphodepleting Conditioning Followed by Infusion of Anti-MART-1 F5 TCR-Gene Engineered Lymphocytes and ALVAC Virus Immunization
Brief Title: Anti-MART-1 F5 Cells Plus ALVAC MART-1 Vaccine to Treat Advanced Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to low accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080056; 08-C-0056
Record Dates: First submitted 2008-02-08; First posted 2008-02-11 (Estimated); Results first posted 2012-04-19 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Metastatic Melanoma; Skin Cancer
Keywords: Immunotherapy; Metastatic Melanoma; Vaccination; Tumor Regression; Skin Cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — aldesleukin; Interleukin-2; Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ALVAC plus anti-MART-1 F5 TCR PBL + HD IL-2 (Experimental): ALVAC plus anti-MART-1 F5 T cell receptor (TCR ) peripheral blood lymphocytes (PBL) + high dose (HD) interleukin 2 (IL-2): ALVAC vaccine-approximately two hours prior to cell infusion, patients will receive 0.5 mL containing a target dose of 10^7 cell culture infectious dose 50% (CCID50) (with a range of approximately 10^6,4 to 10^7,9/mL) of the MART-1 ALVAC virus subcutaneously in each extremity (total of 4 x 10^7 CCID50/2 mL). This will be repeated on day 14.
  Aldesleukin - 720,000 IU/kg intravenously over 15 minutes every 8 hours (+/- 1 hour) for up to 5 days.
  Interventions: Biological: autologous anti-MART-1 F5 T-cell receptor gene-engineered peripheral blood lymphocytes; Biological: ALVAC MART-1 Vaccine; Biological: aldesleukin; Drug: cyclophosphamide; Drug: fludarabine phosphate

INTERVENTIONS:
Biological: autologous anti-MART-1 F5 T-cell receptor gene-engineered peripheral blood lymphocytes — ALVAC vaccine-approximately two hours prior to cell infusion, patients will receive 0.5 mL containing a target dose of 10^7 CCID50 (with a range of approximately 10^6,4 to 10^7,9/mL) of the MART-1 ALVAC virus subcutaneously in each extremity (total of 4 x 10^7 CCID50/2 mL). This will be repeated on day 14.
Biological: ALVAC MART-1 Vaccine — ALVAC vaccine-approximately two hours prior to cell infusion, patients will receive 0.5 mL containing a target dose of 10^7 CCID50 (with a range of approximately 10^6,4 to 10^7,9/mL) of the MART-1 ALVAC virus subcutaneously in each extremity (total of 4 x 10^7 CCID50/2 mL). This will be repeated on day 14.
Biological: aldesleukin — Aldesleukin - 720,000 IU/kg intravenous over 15 minutes every 8 hours beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum 15 doses)
  Other Names: IL2; Proleukin; Recombinant human interleukin 2
Drug: cyclophosphamide — 60 mg/kg day x 2 days intravenous in 250 ml dextrose 5% in water (D5W) with Mesna 15 mg/kg day x 2 days over 1 hour
  Other Names: Cytoxan
Drug: fludarabine phosphate — 25 mg/m^2 day intravenous piggy back over 30 minutes for 5 days
  Other Names: Fludara

SUMMARY:
Background:

* Melanoma antigen recognized by T-cells (MART)-1 is a protein present in melanoma cells.
* An experimental procedure developed for treating patients with melanoma uses the anti-MART-1 F5 gene and a type of virus to make special cells called anti-MART-1 F5 cells that are designed to destroy the patient's tumor. These cells are created in the laboratory using the patient's own tumor cells or blood cells.
* The treatment procedure also uses a vaccine called plaque purified canarypox vector (ALVAC) MART-1, made from a virus that ordinarily infects canaries and is modified to carry a copy of the MART-1 gene. The virus cannot reproduce in mammals, so it cannot cause disease in humans. When the vaccine is injected into a patient, it stimulates cells in the immune system that may increase the efficiency of the anti-MART-1 F5 cells.

Objectives:

-To evaluate the safety and effectiveness of anti-MART-1 F5 and the ALVAC vaccine in treating patients with advanced melanoma.

Eligibility:

-Patients 18 years of age with metastatic melanoma for whom standard treatments have not been effective.

Design:

* Patients undergo scans, x-rays and other tests and leukapheresis to obtain white cells for laboratory treatment.
* Patients have 7 days of chemotherapy to prepare the immune system for receiving the anti-MART-1 F5.
* Patients receive the ALVAC vaccine, anti-MART-1 F5 cells and interleukin-2 (IL-2) (an approved treatment for advanced melanoma). The anti-MART-1 F5 cells are given as an infusion through a vein. The vaccine is given as injections just before the infusion of anti-MART-1 F5 cells and again 2 weeks later. IL-2 is given as a 15-minute infusion every 8 hours for up to 5 days after the cell infusion for a maximum of 15 doses.
* After hospital discharge, patients return to the clinic for periodic follow-up with a physical examination, review of treatment side effects, laboratory tests and scans every 1 to 6 months.

DETAILED DESCRIPTION:
Background:

* We have engineered human PBLs to express an anti-MART-1 T-cell receptor that recognizes an human leukocyte antigens (HLA-A) 0201 restricted epitope derived from the tumor infiltrating lymphocytes (TIL) clone DMF5.
* We constructed a single retroviral vector that contains both alpha and infinity chains and can mediate genetic transfer of this T cell receptor (TCR) with high efficiency without the need to perform any selection.
* In co-cultures with HLA-A 0201 positive melanoma, anti-MART-1 F5 TCR transduced T cells secreted significant amount of interferon (IFN)-(but no significant secretion was observed in control co-cultures with cell lines.
* The anti-MART-1 F5 TCR transduced peripheral blood lymphocytes (PBL) could efficiently kill HLA-A 0201 positive tumors. There was little or no recognition of normal fibroblasts cells.
* This TCR is over 10 times more reactive with melanoma cells than the MART-1 TCR that mediated tumor regression in two patients with metastatic melanoma.
* In this trial we would like to test our hypothesis that the addition of an anti-tumor ALVAC vaccine will result in clinical tumor regression and persistence of the transferred cells (as is the case in murine models).

Objectives:

Primary objectives:

-Determine if the administration of anti-MART-1 F5 TCR -engineered peripheral blood lymphocytes, ALVAC anti-tumor immunization, and aldesleukin to patients following a nonmyeloablative but lymphoid depleting preparative regimen will result in clinical tumor regression in patients with metastatic melanoma.

Secondary objectives:

* Determine the in vivo survival of TCR gene-engineered cells.
* Determine the toxicity profile of this treatment regimen.

Eligibility:

Patients who are HLA-A 0201 positive and 18 years of age or older must have:

* metastatic melanoma;
* previously received and have been a non-responder to or recurred after aldesleukin;
* normal values for basic laboratory values.

Patients may not have:

* concurrent major medical illnesses;
* any form of primary or secondary immunodeficiency;
* severe hypersensitivity to any of the agents used in this study;
* contraindications for high dose aldesleukin administration.
* Design:
* peripheral blood mononuclear cells (PBMC) obtained by leukapheresis (approximately 5 times 10^9 cells) will be cultured in the presence of anti-CD3 (OKT3) and aldesleukin in order to stimulate T-cell growth.
* Transduction is initiated by exposure of approximately 10^8 to 5 X 10^8 cells to retroviral vector supernatant containing the anti-MART-1 F5 TCR genes. These transduced cells will be expanded and tested for their anti-tumor activity.
* Once engineered PBMC are demonstrated to be biologically active according to the strict-criteria outlined in the Certificate of Analysis, patients will receive a nonmyeloablative but lymphocyte depleting preparative regimen consisting of cyclophosphamide and fludarabine followed by intravenous infusion of ex vivo tumor reactive, TCR gene-transduced PBMC plus intravenous (IV) aldesleukin (720,000 IU/kg q8h for a maximum of 15 doses). Approximately 2 hours prior to cell infusion, patients will be immunized with ALVAC virus expressing the tumor antigen. ALVAC immunization will be repeated at 2 weeks.
* Patients will undergo complete evaluation of tumor with physical examination, computed tomography (CT) of the chest, abdomen and pelvis and clinical laboratory evaluation four to six weeks after treatment and then monthly for approximately 3 to 4 months or until off study criteria are met.
* The study will be conducted using a phase II optimal design where initially 21 evaluable patients will be enrolled. If 0 or 1 of the 21 patients experiences a clinical response, then no further patients will be enrolled but if 2 or more of the first 21 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 41 evaluable patients have been enrolled.
* The objective will be to determine if the combination of high dose aldesleukin, lymphocyte depleting chemotherapy, ALVAC immunization and anti-MART-1 F5 TCR-gene engineered lymphocytes is able to be associated with a clinical response rate that can rule out 5 percent (p0=0.05) in favor of a modest 20 percent partial response (PR) plus complete response (CR) rate (p1=0.20).

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Metastatic melanoma with measurable disease.
2. Previously received high dose interleukin-2 (IL-2) and have been either non-responders (progressive disease) or have recurred.
3. Positive for MART-1 by immunohistochemistry (IHC) which will be reviewed by the Laboratory of Pathology at National Cancer Institute (NCI).
4. Tumor infiltrating lymphocytes (TIL) cells not available for treatment on other Surgery Branch protocols.
5. Greater than or equal to 18 years of age.
6. Willing to sign a durable power of attorney.
7. Able to understand and sign the Informed Consent Document.
8. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
9. Life expectancy of greater than three months.
10. Patients of both genders must be willing to practice birth control for four months after receiving the preparative regimen.
11. Patients must be human leukocyte antigens (HLA-A) 0201 positive.
12. Serology:

    * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune -competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
    * Seronegative for hepatitis B antigen and hepatitis C antibody unless antigen negative.
13. Hematology:

    * Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim.
    * White blood cell (WBC) (greater than 3000/mm^3.
    * Platelet count greater than 100,000/mm^3.
    * Hemoglobin greater than 8.0 g/dl.
14. Chemistry:

    * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less or equal to 2.5 times the upper limit of normal.
    * Serum creatinine less than or equal to 1.6 mg/dl.
    * Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
15. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).
16. Six weeks must have elapsed since prior MDX-010 therapy to allow antibody levels to decline.
17. Patients who have previously received MDX-010 or ticilimumab must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
2. Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
3. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
4. Ongoing opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
5. Systemic steroid therapy.
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
7. History of coronary revascularization or ischemic symptoms.
8. Any patient known to have an left ventricular ejection fraction (LVEF) less than or equal to 45 percent.
9. Documented LVEF of less than or equal to 45 percent tested in patients with:

   * Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block.
   * Age greater than or equal to 60 years old.
10. Documented forced expiratory volume in 1 second (FEV1) less than or equal to 60 percent predicted tested in patients with:

    * A prolonged history of cigarette smoking (20 pk/yrs of smoking).
    * Symptoms of respiratory dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kawakami Y, Eliyahu S, Delgado CH, Robbins PF, Rivoltini L, Topalian SL, Miki T, Rosenberg SA. Cloning of the gene coding for a shared human melanoma antigen recognized by autologous T cells infiltrating into tumor. Proc Natl Acad Sci U S A. 1994 Apr 26;91(9):3515-9. doi: 10.1073/pnas.91.9.3515. PMID 8170938
- [Background] Walter EA, Greenberg PD, Gilbert MJ, Finch RJ, Watanabe KS, Thomas ED, Riddell SR. Reconstitution of cellular immunity against cytomegalovirus in recipients of allogeneic bone marrow by transfer of T-cell clones from the donor. N Engl J Med. 1995 Oct 19;333(16):1038-44. doi: 10.1056/NEJM199510193331603. PMID 7675046
- [Background] Kawakami Y, Eliyahu S, Sakaguchi K, Robbins PF, Rivoltini L, Yannelli JR, Appella E, Rosenberg SA. Identification of the immunodominant peptides of the MART-1 human melanoma antigen recognized by the majority of HLA-A2-restricted tumor infiltrating lymphocytes. J Exp Med. 1994 Jul 1;180(1):347-52. doi: 10.1084/jem.180.1.347. PMID 7516411
- See also: Response Evaluation Criteria in Solid Tumors (RECIST) Criteria — http://ctep.cancer.gov/protocolDevelopment/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four participants were enrolled in this study.
Groups:
- ALVAC Plus Anti-MART-1 F5 TCR PBL + HD IL-2: ALVAC plus anti-MART-1 F5 T cell receptor (TCR ) peripheral blood lymphocytes (PBL) + HD IL-2: ALVAC vaccine-approximately two hours prior to cell infusion, patients will receive 0.5 mL containing a target dose of 10^7 CCID50 (with a range of approximately 10^6,4 to 10^7,9/mL) of the MART-1 ALVAC virus subcutaneously in each extremity (total of 4 x 10^7 CCID50/2 mL). This will be repeated on day 14.
  Aldesleukin (IL2, Proleukin, Recombinant human interleukin 2)- 720,000 IU/kg intravenously over 15 minutes every 8 hours (+/- 1 hour) for up to 5 days.
Period: Overall Study
Arm/Group | ALVAC Plus Anti-MART-1 F5 TCR PBL + HD IL-2
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ALVAC Plus Anti-MART-1 F5 TCR PBL + HD IL-2
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Metastatic Melanoma Who Develop Clinical Tumor Regression (CR or PR)
Description: Clinical tumor response is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v.1.0 criteria. Complete response (CR) is a disappearance of all target lesions. Partial response (PR) is a 30% decrease in lesions taking as reference the baseline sum longest diameter (LD). For details about the RECIST criteria see the protocol link module.
Time Frame: 4-6 weeks after treatment and then monthly for approximately 3 to 4 months or until off study criteria are met
Measure: Number; unit: Participants
Arm/Group | ALVAC Plus Anti-MART-1 F5 TCR PBL + HD IL-2
Number analyzed (Participants) | 4
Participants | 0

2. Secondary Outcome: Number of Participants With in Vivo Survival of T-cell Receptor (TCR) Gene-engineered Cells
Description: T cell receptor (TCR) and vector presence will be quantitated in peripheral blood mononuclear cells (PBMC) samples using established polymerase chain reaction (PCR) techniques. This will provide data to estimate the in vivo survival of lymphocytes derived from the infused cells.
Time Frame: 1 month
Population: This outcome measure was not done because the study was terminated due to low accrual.
Arm/Group | ALVAC Plus Anti-MART-1 F5 TCR PBL + HD IL-2
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 15 months
Measure: Number; unit: Participants
Arm/Group | ALVAC Plus Anti-MART-1 F5 TCR PBL + HD IL-2
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | ALVAC Plus Anti-MART-1 F5 TCR PBL + HD IL-2
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALVAC Plus Anti-MART-1 F5 TCR PBL + HD IL-2 (N=4)
Hearing test abnormal (Ear and labyrinth disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALVAC Plus Anti-MART-1 F5 TCR PBL + HD IL-2 (N=4)
Hearing test abnormal (Ear and labyrinth disorders) | 1 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 4 (4)
Leukocyte count decreased (Blood and lymphatic system disorders) | 4 (4)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 4 (6)
Neutrophil count decreased (Blood and lymphatic system disorders) | 4 (4)
Platelet count decreased (Blood and lymphatic system disorders) | 4 (4)
Hypotension (Vascular disorders) | 1 (1)
Activated partial thromboplastin time prolonged (aPTT) (Investigations) | 1 (1)
Fatigue (General disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2)
Febrile neutropenia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Catheter-related infection (Infections and infestations) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2)
Bilirubin increased (Metabolism and nutrition disorders) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (2)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Psychosis (Nervous system disorders) | 1 (1)
Speech disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No